CLINICAL TRIAL: NCT02166671
Title: Humoral and Cellular Immune Responses to a Hepatitis B Vaccine Booster 20-23 Years After Neonatal Immunization
Brief Title: Immune Response to Hepatitis B Virus Booster Vaccination After 20-23 Years
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants were not recruited promptly
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HBV_VAX_DUR_2014
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis B Vaccination

ARMS (1):
- HBV booster vaccination (Experimental)
  Interventions: Biological: HBV booster vaccination 1dose

INTERVENTIONS:
Biological: HBV booster vaccination 1dose

SUMMARY:
This study will evaluate the humoral and cellular immune responses to a hepatitis B vaccine booster in healthy adults which received a full course of neonatal hepatitis B vaccination 20-23 years ago.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 20-25 years old

Exclusion Criteria:

* Hepatitis B surface antigen (+)
* Hepatitis B core antibody (+)
* any history of liver disorders including hepatitis
* HIV Ag or Ab(+)

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
change of HBsAb titer | 28 days after HBV booster vaccination

SECONDARY OUTCOMES:
HBsAg-specific cell mediated immunity | 28 days after HBV booster vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea